CLINICAL TRIAL: NCT01063998
Title: A Urinary Tumor Marker (Kidney Injury Molecule-1) for the Detection of Renal Cell Carcinoma
Status: Terminated | Type: Observational
Why Stopped: Preliminary data did not show expected outcomes.
Sponsor: Jason Hafron (Other)
Collaborators: Corewell Health East (Other)
Responsible Party: Sponsor-Investigator, Jason Hafron, Chairman, Dept of Urology, Corewell Health East
Organization: Corewell Health East (Other)
Other Study IDs: 2009-125
Record Dates: First submitted 2009-09-02; First posted 2010-02-05 (Estimated); Last update posted 2013-11-08 (Estimated); Status verified 2013-11

CONDITIONS: Renal Cell Carcinoma
Keywords: Renal cell; Carcinoma; Biomarkers
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Renal tumor.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Patients demonstrate normal serum creatinine and no radiological evidence of a renal tumor.
  Interventions: Other: Urine Marker
- p 2: Patients diagnosed with renal cancer and normal creatinine.
  Interventions: Other: Urine Marker

INTERVENTIONS:
Other: Urine Marker — Urinary KIM-1 measurements
  Other Names: Urine biomarkers; KIM-1

SUMMARY:
The ultimate goal of this project is to develop a simple non-invasive method to screen patients for potential kidney tumors.

DETAILED DESCRIPTION:
In the United States there were 38,900 cases and 12,840 deaths from renal cell carcinoma in 2006. Renal cell carcinoma represents 2% of all cancers worldwide. The majority of kidney tumors are discovered incidentally during investigation of unrelated complaints. However, nearly 30% of patients present with metastatic disease at the time of diagnosis and 30-40% of patients with clinically localized kidney cancer will have a recurrence. The diagnosis and monitoring of kidney cancer requires expensive and frequent imaging examinations. There is a significant need to find diagnostic and prognostic biomarkers to screen, diagnose, and monitor renal cancers.

A reliable urinary assay for kidney cancer would have major implications for tumor screening in high risk patients, in selection of patients for adjuvant therapy, in surveillance and prognosis and possibly as a surrogate marker for response to therapy. Human kidney injury molecule-1 (KIM-1) has been found to be a sensitive and specific biomarker in identifying kidney injury. The urine levels of KIM-1 are increased in the patients with kidney failure and major types of kidney tumors. The purpose of the study is investigate how urine KIM-1 and a routine blood marker for renal failure (creatinine) can distinguish kidney tumors from non-tumor kidney injury. The ultimate goal of this project is to develop a simple non-invasive method to screen patients for potential kidney tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients demonstrate normal serum creatinine and no radiological evidence of a renal tumor.

OR

* Patients diagnosed with renal cancer and normal creatinine.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having nephrectomy.
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To test the sensitivity and specificity of KIM-1 urine excretion in a group of patients with kidney cancer. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hafron, MD, Principal Investigator — Beaumont Hospitals
Locations (1):
- Beaumont Hospitals, Royal Oak, Michigan, United States